CLINICAL TRIAL: NCT00694681
Title: Enhanced Services for the Hard to Employ Demonstration: Telephonic Care Management for Depressed Medicaid Recipients
Brief Title: Working Toward Wellness
Acronym: WtW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDRC (Other)
Collaborators: United Behavioral Health (Industry); Kaiser Permanente (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Michalopoulos, Chief Economist, MDRC
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HHS-233-01-0012-RI
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: Telephonic care management
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Telephonic care management — Individuals received intensive outreach from care managers, first to help them to enter treatment and then, if treatment began, to remain in it for an appropriate time. Treatment is based on the American Psychiatric Association's Evidence-Based Practice Guidelines for Major Depression, which includes psychotherapy and antidepressant medications. Outreach and care management took place by telephone.

SUMMARY:
Working toward Wellness is a telephone care management and outreach monitoring program designed to help Medicaid recipients who are experiencing major depression to enter and remain in evidence-based treatment. To study the effects of Working toward Wellness, individuals receiving Medicaid in Rhode Island who are eligible for mental health services through United Behavioral Health were screened by telephone for depression. Those who were found to have major depression and who agreed to be in the study were randomly assigned. Program participants received intensive monitoring from Master's level clinicians called care managers to facilitate and support clinical treatment. The control group received usual care that included only referrals to mental health treatment providers. The study hypothesis is that telephonic care management would increase visits to mental health professionals and use of appropriate medication, which in turn would reduce depression severity and lead to greater employment and productivity at work.

ELIGIBILITY:
Inclusion Criteria:

* Score of 5 or higher on Quick Inventory of Depression Symptomatology
* receiving Medicaid
* at least one child in household

Exclusion Criteria:

* Bipolar disorder
* alcohol or substance abuse
* currently in active treatment for depression
* receiving Supplemental Security Income

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2004-10; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Use of mental health services | Through 36 months

SECONDARY OUTCOMES:
Depression severity | 6, 18, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: David Butler, Principal Investigator — MDRC
Locations (1):
- United Behavioral Health, Warwick, Rhode Island, United States

REFERENCES:
- [Result] Kim SE, Le Blanc AJ, Michalopoulos C, Azocar F, Ludman EJ, Butler DM, Simon GE. Does telephone care management help Medicaid beneficiaries with depression? Am J Manag Care. 2011 Oct 1;17(10):e375-82. PMID 21999717
- [Result] Kim S, Leblanc A, Morris P, Simon G, Walter J. Working toward wellness: Telephone care management for Medicaid recipients with depression, thirty-six months after random assignment. New York: MDRC. December 2011.